CLINICAL TRIAL: NCT07090304
Title: China Colorectal Cancer Screening Trial 2 (C-Cost2): FIT Versus FIT-sDNA in the Average Risk Population
Brief Title: China Colorectal Cancer Screening Trial 2 (C-Cost2)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Ding Ke-Feng, Professor, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: C-Cost2
Record Dates: First submitted 2025-07-20; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Colorectal Cancer; Advanced Adenoma
Keywords: FIT; FIT-sDNA; Colorectal cancer; Advanced colorectal adenoma; Early screening; Average risk population
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FIT group (Active Comparator): The internationally recommended screening protocol is adopted. In the first 4 years of the screening phase, all participants will receive annual FIT tests. Participants with positive FIT results are recommended to undergo diagnostic colonoscopy. Suspicious lesions detected during the colonoscopy will be resected and further sent for pathological examination. Participants who refuse FIT tests, have negative FIT tests, have positive FIT tests but do not receive diagnostic colonoscopy will be screened again in the first 4 years. All the participants will be followed by long-term follow-ups.
  Interventions: Diagnostic Test: FIT
- FIT-sDNA group (Experimental): A new screening protocol is adopted. In the first 4 years of the screening phase, all participants will receive annual FIT-sDNA tests. Participants with positive FIT-sDNA results are recommended to undergo diagnostic colonoscopy. Suspicious lesions detected during the colonoscopy will be resected and further sent for pathological examination. Participants who refuse FIT-sDNA tests, have negative FIT-sDNA tests, have positive FIT-sDNA tests but do not receive diagnostic colonoscopy will be screened again in the first 4 years. All the participants will be followed by long-term follow-ups.
  Interventions: Diagnostic Test: FIT-sDNA

INTERVENTIONS:
Diagnostic Test: FIT — FIT stands for Fecal Immunochemical Test, a non-invasive screening tool used primarily to detect hidden blood in the stool, which may indicate colorectal cancer or precancerous polyps. Positive cut-off level: 100 ng/mL.
  Arms: FIT group
Diagnostic Test: FIT-sDNA — FIT-sDNA test combines Fecal Immunochemical Test (FIT) and stool DNA (sDNA) analysis. It detects hemoglobin in stool through FIT to identify occult blood in the gastrointestinal tract and simultaneously analyzes specific DNA mutations or epigenetic alterations (such as methylation changes) in stool DNA to assess the risk of colorectal neoplasms.
  Arms: FIT-sDNA group

SUMMARY:
Colorectal cancer (CRC) is one of the most common malignancies in China. Currently, its incidence rate is increasing at a rate of 4% per year, exceeding the global annual average growth rate. Screening and early diagnosis of colorectal cancer and precancerous lesions are key measures to reduce the disease burden of colorectal cancer in China. In previous clinical studies, colorectal cancer screening in high risk population received extensive attention. However, it cannot be ignored that the majority of sporadic colorectal cancers occur in the average risk population. Therefore, there is an urgent need to develop new approach for colorectal cancer screening in the average risk population in China.

Fecal Immunochemical Testing (FIT) initial screening followed by diagnostic colonoscopy is widely recommended by colorectal cancer screening guidelines worldwide. The current colorectal cancer screening approach faces challenges including limited sensitivity of initial screening technologies and insufficient population coverage in organized screening programs in China. Stool DNA tests detect DNA biomarkers of tumor cells in the stool and have higher sensitivity in detecting advanced colorectal neoplasms. USPSTF has recommended FIT-sDNA as initial screening tests in the average risk population. Colorectal Cancer Early Screening in China (Clear-C) trial has reported FIT-sDNA had higher sensitivity than FIT in detecting advanced colorectal neoplasms among high risk population, yet there is a lack of randomized controlled trials (RCTs) directly comparing the effectiveness of FIT and FIT-sDNA for colorectal cancer screening in the average risk population in China.

In China Colorectal Cancer Screening Trial 2 (C-Cost2), we propose to perform a multicenter, individual-level randomized, parallel group trial directly comparing FIT and FIT-sDNA in the average risk population in China. The main research hypothesis is that the screening protocol of FIT-sDNA group (Group B) has a superior detection rate of advanced colorectal neoplasms compared to the FIT group (Group A).

DETAILED DESCRIPTION:
This study intends to recruit participants who meet the above inclusion and exclusion criteria in China, with the goal of recruiting at least 7504 eligible participants at baseline. The study adopts an individual-level randomized design. After signing the informed consent form, eligible participants will be randomly assigned to 2 colorectal cancer screening groups. All participants will undergo a 4-year screening phase, and then all participants will be followed up for a long term. Fecal, blood, and tissue samples will be collected from the participants during the study. The grouping and specific intervention measures are as follows:

1. FIT group (n = 3752): The internationally recommended screening protocol is adopted. In the first 4 years of the screening phase, all participants will receive annual FIT tests. Participants with positive FIT results are recommended to undergo diagnostic colonoscopy. Suspicious lesions detected during the colonoscopy will be resected and further sent for pathological examination. Participants who refuse FIT tests, have negative FIT tests, have positive FIT tests but do not receive diagnostic colonoscopy will be screened again in the first 4 years. All the participants will be followed by long-term follow-ups.
2. FIT-sDNA group (n = 3752): A new screening protocol is adopted. In the first 4 years of the screening phase, all participants will receive annual FIT-sDNA tests. Participants with positive FIT-sDNA results are recommended to undergo diagnostic colonoscopy. Suspicious lesions detected during the colonoscopy will be resected and further sent for pathological examination. Participants who refuse FIT-sDNA tests, have negative FIT-sDNA tests, have positive FIT-sDNA tests but do not receive diagnostic colonoscopy will be screened again in the first 4 years. All the participants will be followed by long-term follow-ups.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 45-74 years old;
2. In good general condition, with normal mental state and voluntarily signing the informed consent form;

Exclusion Criteria:

1. Personal history of colorectal cancer or precancerous lesions;
2. History of previous colonrectal resection surgery;
3. Diagnosed with cancer before enrollment or currently receiving any cancer-related treatment;
4. Having received colonoscopy, flexible sigmoidoscopy, CT colonography and other examinations within the past 5 years;
5. Having received FIT or FIT-sDNA or cfDNA test within the past 1 year;
6. Symptomatic lower gastrointestinal diseases or symptoms suggesting the need for diagnostic colonoscopy for confirmation;
7. Accompanied by severe diseases that are not suitable for colorectal cancer screening;

Ages: 45 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7504 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Detection rate of advanced colorectal neoplasms | 4 years
  Advanced colorectal neoplasms includes advanced adenomas and colorectal cancer

SECONDARY OUTCOMES:
Population compliance rate | 4 years
  Population compliance rate
Proportion of colorectal cancer at different stages | 4 years
  Proportion of colorectal cancer at different stages
Incidence rate of colorectal cancer | 10 years
  Incidence rate of colorectal cancer
Mortality rate of colorectal cancer | 10 years
  Mortality rate of colorectal cancer
Quality of life (QOL) | 4 years
  Quality of life will be assessed by EuroQol five-dimensional questionnaire (EQ-5D）
Total cost and cost per detected lesion | 4 years
  Total cost and cost per detected lesion
Incremental cost-effectiveness ratio | 4 years
  Incremental cost-effectiveness ratio

IPD SHARING:
Plan to Share IPD: No